CLINICAL TRIAL: NCT03069872
Title: Access to Fast Transvaginal Ultrasound Through General Practice for Earlier Diagnosis of Ovarian Cancer
Brief Title: A Trial of Fast Access to Transvaginal Ultrasound Through General Practice for Earlier Diagnosis of Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 210278
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2018-04

CONDITIONS: Ovarian Cancer
Keywords: Transvaginal ultrasound; General practice; Early diagnosis; Symptoms
MeSH Terms: conditions — Ovarian Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All GPs in Central Denmark Region, are planned to be enrolled in the study during the one year study period.
  Interventions: Diagnostic Test: Transvaginal ultrasound

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound — Access to fast transvaginal ultrasound through general practice Develop and conduct training for general practicioners in the latest knowledge of ovarian cancer symptomatology

SUMMARY:
Background

Ovarian cancer (OC) is a disease with a poor prognosis due to diagnosis at late stage. Early-stage OC presents with non-specific and vague symptoms and therefore OC usually is not detected until reaching an advanced stage. From 2008, Danish general practitioners (GPs) could urgently refer patients suspected of having OC to standardized cancer patient pathways (CPPs). The CPP is designed for women presenting specific signs and alarm symptoms, and is supposed to shorten the pathway from suspicion to treatment.

Hypothesis

Direct access to fast transvaginal ultrasound (TVU) through general practice is feasible in earlier diagnosis of OC.

Aim

The aim of this study is to assess the implementation and clinical implications of direct referral access to fast TVU through general practice.

Materials and methods

The study is a feasibility study and GPs from in Central Denmark Region are offered direct access to fast TVU for women aged 40 years or more who present symptoms that could origin from OC, but which are not classified as alarm symptoms. The GPs will receive education about updated knowledge on OC symptoms and the use of the guideline for earlier diagnosis of OC in general practice. The study period is 1 year.

Perspectives

There is a great need to test rational strategies for diagnosing OC at an earlier stage in order to improve survival. For women who do not fulfil access criteria for the CPP, and for whom the main prospect for earlier diagnosis is improved identification of symptomatic OC, this study may provide important new knowledge of how to facilitate the diagnostics of OC in the future and reduce time to diagnosis and improve survival.

DETAILED DESCRIPTION:
Background

Around 550 ovarian cancers (OCs) are diagnosed yearly in Denmark. Still, OC is the fourth commonest cause of cancer death amongst women in Denmark. Epithelial ovarian cancers (carcinomas) account for more than 90% of all OCs and Denmark has the second highest incidence in the world (15 per 100.000 women) with a life-time risk around 2%. The mean age at diagnosis is 63 years, and 80% are postmenopausal. In Denmark, 74% are diagnosed in FIGO stage III-IV and therefore at the time of diagnosis have regional or metastatic spread. Five-year survival with FIGO stage I is 83%, stage II 62%, stage III 23% and stage IV 11%. Thus, OC is detected at advanced stages with a very poor prognosis.

In 2008, a national fast-track system for cancer patients was established to ensure fast diagnosis and initiation of treatment. The fast-track system or cancer patient pathway (CPP) implies that patients presenting 'alarm' symptoms of e.g. OC will be referred immediately for diagnostic workup; no more than 14 days must pass from referral to initiation of treatment. Only about one quarter of the women with OC are referred primarily through this route. Therefore, additional accelerated routes are needed for the majority of women with OC.

A possibility could be access to fast TVU through general practice for women presenting with vague and non-specific symptoms that may represent underlying OC.

Aim

Develop and conduct training for general practitioners (GPs) in the latest knowledge of OC symptomatology. And at the same time investigate the feasibility and clinical implications in general practice of direct referral access to fast TVU, intended for women presenting with vague and non-specific symptoms.

Material and methods

GPs in Central Denmark Region are offered direct access to fast TVU for women aged 40 years or more who present vague and non-specific symptoms that could origin from OC, but which are not classified as alarm symptoms. Shortly afterwards all the GPs are offered a short lecture on OC symptomatology and instructions for the use of TVU for earlier diagnosis of OC through general practice. The lecture will be conducted by researchers from the research group.

Prior to investigation, all women who are referred to TVU will receive a consent form and a symptom-questionnaire. The symptom questionnaire focuses on the experienced symptoms during the past year.

After finished investigation, the TVU test results will return electronically to the referring GP.

The study period is one year. Data analysis will focus on the frequency of TVU use in general practice, action taken on test results and patient-reported symptoms prior to TVU.

Perspectives

The project will provide important new knowledge of the GPs referral practice when they suspect OC. For women presenting with vague and non-specific symptoms that may origin from OC, the introduction of TVU through general practice will provide new possibilities for evaluating the symptoms. Therefor introduction of TVU is a corner stone in the identification of more efficient ways to evaluate women at risk of developing OC.

This study will contribute with important knowledge of how to improve the diagnostics of OC in the future and may reduce time to diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* GPs in the Central Denmark Region
* Women ≥40 years presenting with vague and non-specific symptoms

Exclusion Criteria:

* Women who fulfil access criteria for OC fast-track referral.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Frequency of TVU use | one year
  TVU will be requested electronically through an online referral-system used by Danish GPs.
  This outcome will be evaluated descriptively by illustrating the relation between time and use of TVU.
Action taken on test results | one year
  After all TVU investigations, a discharge summary will be send electronically to the referring GP.
  If indicated, instructions for follow-up investigations is stated in the discharge summary. To evaluate if GPs follow these instructions, data on discharge summary recommended follow-up are compared to data on follow-up referrals made by the GPs. This outcome will be evaluated descriptively.
Patient-reported symptoms before TVU investigation | one year
  All women who are referred to TVU will receive a questionnaire prior to investigation, regarding experienced symptoms during the past year.
Indication for fast TVU | one year
  GPs refer women to TVU electronically. Information about indications for the investigation, is required in the referral. These informations will be used to evaluate the GPs reasons for referring the women to TVU and will be evaluated descriptively.

SECONDARY OUTCOMES:
Findings by TVU on women with vague and non-specific symptoms | one year
  An overview of all findings by TVU will be provided, and possible side effects will be assessed.
  An algorithm for the use of TVU has been developed, and the principal investigator will tick a box specifying what has been discovered during the investigation. Findings by TVU is identified in the algorithm used for TVU and by ICD-10 codes.
Ovarian Cancer (OC) stage distribution | one year
  Number of OC diagnosed in each cancer stage (FIGO I-IV)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Louise L Baun, MD, Principal Investigator — Research Unit of General Practice, Aarhus University; Peter Vedsted, Professor, Study Director — Research Unit of General Practice, Aarhus University; Margit Dueholm, As.Professor, Study Chair — Aarhus University Hospital; Lone Kjeld Petersen, As.Professor, Study Chair — Department of Gynaecology, Randers Regional Hospital
Locations (1):
- Aarhus University, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No